CLINICAL TRIAL: NCT01976637
Title: Compression Treatment of Superficial Vein Thrombosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Kornelia Boehler, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EKNr 772/2009
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Pain; Erythema; Thrombus Length; Quality of Life
MeSH Terms: conditions — Pain; Erythema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- no compression (Experimental): no compression stockings worn during a 3 weeks period
  Interventions: Other: no compression
- compression stockings (Active Comparator): compression stockings class II (23-32 mm Hg) worn during the day for up to 3 weeks
  Interventions: Device: compression

INTERVENTIONS:
Other: no compression — no compression stockings worn during the study
  Arms: no compression
Device: compression — compression stockings class II (23-32 mm Hg) worn during the day for up to 3 weeks
  Arms: compression stockings

SUMMARY:
Leg compression is considered the basic treatment for superficial vein thrombosis (SVT). However, its use is more or less based on subjective experience while scientific evidence for its efficacy is lacking. There is one uncontrolled trial reporting improvement of clinical symptoms when patients with SVT were treated with fixed compression bandages.

This study evaluates the efficacy of compression stockings (23-32 mmHg) in the treatment SVT of the legs. The investigators hypothesis is that compression treatment is superior to no compression in alleviating disease related clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* patients with superficial vein thrombosis of the leg,
* thrombus extent of at least 5 cm confirmed by duplex sonography,
* clinical signs of inflammation (pain, erythema)

Exclusion Criteria:

* superficial thrombus distance to the saphenofemoral or saphenopopliteal junction of less than 2cm,
* concomitant deep vein thrombosis,
* thrombophilia,
* active malignoma,
* immobility,
* peripheral arterial occlusive disease,
* superficial vein thrombosis after sclerotherapy
* incision and clot expression
* excessive leg configuration not covered by ready made compression stockings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
pain assessed by VAS (cm) | at baseline, week 1, week 2, week 3
  change from baseline to week 3 at weekly intervals

SECONDARY OUTCOMES:
skin erythema (cm2) | at baseline, week 1, week 2, week 3
  change from baseline to week 3 at weekly intervals
duplex-sonographic change in thrombus length (cm) | at baseline, week 1, week 2, week 3
  change from baseline to week 3 at weekly intervals
quality of life (SF-36) | at baseline and at week 3
  change from baseline to week 3
amount of analgetics (number of pills) | week 1, week 2, week 3
  change from week 1 to week 3
duplex-sonographic confirmation of deep vein thrombosis | at baseline and at week 3
löwenberg test (mm Hg) | at baseline, week 1, week 2, week 3
  change from baseline to week 3

OTHER OUTCOMES:
D-dimer ug/ml | at baseline and at week 3
platelet count | at baseline, day 7 and day14

CONTACTS AND LOCATIONS:
Overall Officials: Kornelia Böhler, MD, Principal Investigator — Medical University of Vienna, Department of General Dermatology